CLINICAL TRIAL: NCT06019858
Title: A Clinical Trial to Assess the Effects of a Vitamin Shot on Energy Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitamin Energy® (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20348
Record Dates: First submitted 2023-08-24; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Energy; Fatigue; Mood; Weight Loss; Cognition
MeSH Terms: conditions — Fatigue; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitamin Energy Shot (Experimental): Participants will take one bottle daily of the Vitamin Energy® shot, in the morning.
  Interventions: Other: Vitamin Energy Shot

INTERVENTIONS:
Other: Vitamin Energy Shot — Vitamin Energy® shot is a naturally-caffeinated functional energy shot that contains:
  Vitamin B3 Vitamin B6 Vitamin B12 Natural Caffeine (green tea extract) L-Carnitine Tartrate Potassium Sorbate Taurine Sucralose

SUMMARY:
This is a virtual, single-arm clinical trial that will last 30 days. Participants will drink 1 bottle of the Vitamin Energy® shot daily and complete questionnaires at baseline, Day 7, Day 14, and Day 30.

Participants' energy, mood, and cognitive function will be evaluated at baseline and at each check-in. Bodyweight will also be assessed at baseline and Day 30. Likert scale responses will be examined from baseline to each check-in. Participant responses on product feedback will be presented as % scores.

ELIGIBILITY:
Inclusion Criteria:

Men and women 18 years and over

Self-reported issues with:

* Energy
* Focus
* Brain fog Participants who often feel fatigued Willing to maintain the same caffeine consumption during the study period Generally healthy - don't live with any uncontrolled chronic disease

Exclusion Criteria:

Any pre-existing chronic conditions that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders.

Anyone with known severe allergic reactions. Women who are pregnant, breastfeeding, or attempting to become pregnant Unwilling to follow the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-06-21 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Change in energy levels. [Baseline to Day 30] | 30 days
  Survey-based assessment (0-5 scale) of participant reported energy levels.

SECONDARY OUTCOMES:
Change in ability to concentration. [Baseline to Day 30] | 30 days
  Survey-based assessment (0-5 scale) of participant reported concentration abilities.
Change in participant-perceived productivity. [Baseline to Day 30] | 30 days
  Survey-based assessment (0-5 scale) of participants perception of their productivity during the day.
Changes in mood. [Baseline to Day 30] | 30 days
  Survey-based assessment (0-5 scale) of mood.
Changes in brain fog. [Baseline to Day 30] | 30 days
  Survey-based assessment (0-5 scale) of brain fog experienced by participants.
Change in body weight. [Baseline to Day 30] | 30 days
  Participants will weight themselves at baseline and endline and provide their body weight.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided